CLINICAL TRIAL: NCT07407244
Title: Study AKRA: Correlation of Immune-Related Tumor Stroma Factors With Complete Pathologic Remission in Early Breast Cancer After Neoadjuvant Chemotherapy and With Circulating Tumor Cells/Circulating Tumor DNA
Brief Title: Immune Tumor Stroma Factors and Pathologic Complete Response After Neoadjuvant Chemotherapy in Early Breast Cancer
Acronym: AKRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OIL_AKRA _EBC; P3-0321 (Other: ARIS (Slovenian Research and Innovation Agency))
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemotherapy for Early Breast Cancer (Other): Patients with early breast cancer receiving standard neoadjuvant chemotherapy will be followed to assess immune-related tumor stroma factors and blood biomarkers in association with complete pathologic remission (pCR) and circulating tumor cells/circulating tumor DNA.
  Interventions: Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Standard neoadjuvant chemotherapy administered to patients with early breast cancer according to institutional protocols. Treatment is not experimental and is part of routine clinical care. Immune-related tumor stroma factors and blood biomarkers will be analyzed in relation to pathological complete response (pCR) and circulating tumor cells/circulating tumor DNA.

SUMMARY:
This prospective cohort study aims to identify immune-related predictive factors of response to neoadjuvant chemotherapy in patients with early breast cancer. The study will evaluate immune markers in tumor stroma and blood samples collected before treatment to determine their association with complete pathological remission (pCR). In addition, circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) will be analyzed to explore their correlation with treatment response. The results may contribute to improved selection of patients who are most likely to benefit from neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This prospective observational cohort study investigates the relationship between immune-related tumor stroma factors and response to neoadjuvant chemotherapy (NACT) in patients with early breast cancer treated at the Institute of Oncology Ljubljana.

The primary objective is to identify immune predictive markers in the tumor microenvironment that are associated with achieving pathological complete remission (pCR) after neoadjuvant chemotherapy. Tumor tissue and blood samples will be analyzed to evaluate immune-related biomarkers and their prognostic and predictive value.

In addition, circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA) will be assessed in peripheral blood samples collected before initiation of treatment, in order to determine their association with immune-related tumor stroma characteristics and clinical outcomes.

The study aims to improve understanding of biological mechanisms influencing treatment response and may support future personalized treatment strategies by identifying patients who are most likely to benefit from neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Female patients with early breast cancer

Planned neoadjuvant chemotherapy (NACT)

Availability of tumor tissue sample (biopsy) before treatment

Ability to provide blood sample(s)

Signed informed consent

Exclusion Criteria:

Male breast cancer

Patients without neoadjuvant chemotherapy

Inability or refusal to provide informed consent

Insufficient biological material for analysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | After completion of neoadjuvant chemotherapy (at surgery)
  To determine immune-related predictive factors of response to neoadjuvant chemotherapy in the tumor stroma of patients with early breast cancer, in relation to achieving pathological complete response (pCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No